CLINICAL TRIAL: NCT01811160
Title: Metabolic Effects of Melatonin in Patients Treated With Second Generation Antipsychotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Responsible Party: Principal Investigator, Francisco Romo Nava, MD, Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INPRF_144; INPRF_144 (Other Grant/Funding Number: Instituto Nacional de Psiquiatría No. 144)
Record Dates: First submitted 2013-02-28; First posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Second Generation Antipsychotic Induced Metabolic Adverse Effects
Keywords: Melatonin; Second generation antipsychotic; bipolar disorder; schizophrenia; Metabolic
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin 5mg (extended release capsules) (Experimental): Subjects received melatonin (extended release) 5mg nightly during the follow up period
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Subjects received a placebo capsule nightly during the eight week follow up period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — A capsule of melatonin was administered nightly (20:00hrs).
  Other Names: Melatonin 5mg capsules were administered at 20:00hrs during the follow up period.
  Arms: Melatonin 5mg (extended release capsules)
Drug: Placebo — Placebo capsules were administered at 20:00hrs for eight weeks
  Arms: Placebo

SUMMARY:
Schizophrenia and bipolar disorder are frequently associated with an elevated risk for obesity, metabolic syndrome, diabetes mellitus, dyslipidemia and other metabolic disturbances. Second Generation Antipsychotics (SGA) have a demonstrated efficacy in acute and long term treatment of these disorders and are considered a first option on most treatment guidelines. Unfortunately the use of SGA is associated to drug induced weight gain, disturbed glucose and lipid regulation and an increase of cardiovascular risk and mortality as well as non- adherence to treatment. There are several hypotheses attempting to explain the complex pathways that lead to antipsychotic therapeutic effects and their accompanying adverse effects. Recently, in animals receiving SGA, melatonin prevented to a large extent the body weight increase, which indicates a possible role for biological rhythms in SGA induced body weight accumulation. Melatonin is a hormone secreted by the pineal gland that follows a circadian rhythm with an increased secretion in the middle of the night. This hormone acts importantly on the suprachiasmatic nucleus and other areas in the brain and periphery. Thus melatonin is involved in a series of biological functions such as sleep regulation, blood pressure, regulation of circadian rhythms, mood, behavior, and more recently in the regulation of metabolic processes including insulin, leptin, and lipid regulation.

Given previous results in experimental animals, the purpose of the present study is to test the potential effect of melatonin in reducing or preventing some of the metabolic disturbances associated with SGA

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant, non-lactating women aged between 18 and 45 years;
2. DSM-IV-TR criteria for schizophrenia or bipolar disorder type I;
3. free of concomitant medical or neurological illness (as per review of systems and general physical examination);
4. free of DSM-IV current substance abuse or a history of substance dependence in the last six months;
5. who were initiated on continuous treatment with SGA (clozapine, olanzapine, quetiapine or risperidone) for a period no greater than the last three months prior to their inclusion to the present study.

Exclusion Criteria:

1. were diagnosed with hypertension, diabetes mellitus, dyslipidemia, thyroid disorders or hepatic illness;
2. had a history of hypersensitivity to melatonin;
3. exhibited high risk for suicide or high risk for aggressiveness;
4. women who were not practicing reliable forms of contraception. Patients were eliminated from the study if they suspended SGA or two consecutive doses of the study capsule at any point during the follow up period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Weight change | Mean change from baseline weight at 8 weeks

SECONDARY OUTCOMES:
Mean change in systolic blood pressure | Mean change from baseline systolic blood pressure at 8 weeks
Mean change diastolic blood pressure | Mean change from baseline diastolic blood pressure at 8 weeks
Mean change waist circumference | Mean change from baseline waist circumference at 8 weeks
Mean change hip circumference | Mean change from baseline hip circumference at 8 weeks
Mean change fat mass | Mean change from baseline fat mass at 8 weeks
Mean change lean mass | Mean change from baseline lean mass at 8 weeks
Mean change total body water | Mean change from baseline total body water at 8 weeks
Mean change glucose | Mean change from baseline glucose at 8 weeks
Mean change low density lipoprotein | Mean change from baseline low density lipoprotein at 8 weeks
Mean change high density lipoprotein | Mean change from baseline high density lipoprotein at 8 weeks
Mean change triglycerides | Mean change from baseline triglycerides at 8 weeks
Mean change cholesterol | Mean change from baseline cholesterol at 8 weeks
Mean change Hamilton D scores | Mean change from baseline Hamilton D score at 8 weeks
Mean change Young Mania rating scale | Mean change from baseline Young Mania rating scale at 8 weeks
Mean change Positive and Negative Symptoms scale | Mean change from baseline Positive and Negative Symptoms scale at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Romo-Nava, MD, Principal Investigator — Instituto Nacional de Psiquiatría / UNAM
Locations (1):
- Instituto Nacional de Psiquiatría "Dr. Ramón de la Fuente", Mexico City, México City, Mexico